CLINICAL TRIAL: NCT06964880
Title: The Effectiveness of a Media Integration Peer Support Model in Enhancing Awareness and Health Behaviors Related to Obesity and Sarcopenic Obesity Among Overweight-risk College Students
Brief Title: Effectiveness of a Peer Support Media Model on Obesity and Sarcopenia Awareness in At-Risk College Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CMUH113-REC1-164
Record Dates: First submitted 2025-03-04; First posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Exercise Adherence
Keywords: Sarcopenic obesity; body fat percentage; muscle mass; exercise; audiovisual media
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online Video Exercise + Peer Support (Experimental): Participants in the intervention group will engage in a 12-week program that includes twice-weekly structured exercise sessions guided by video content delivered via an online media platform. The program also includes weekly health education videos on nutrition and sarcopenic obesity. Participants will be organized into peer support groups (5 members per group) to promote mutual encouragement and accountability in maintaining healthy behaviors.
  Interventions: Behavioral: Exercise with video on media platform
- Printed Health Education Materials (Active Comparator): Participants in the control group will receive printed health education materials weekly for 12 weeks. These materials cover the same topics as the intervention group, including healthy eating, physical activity, and prevention of sarcopenic obesity, but without the video-based guidance or peer group support.
  Interventions: Behavioral: Printed Educational Handout

INTERVENTIONS:
Behavioral: Exercise with video on media platform — 12-week structured video-guided exercise and peer support program
  Arms: Online Video Exercise + Peer Support
Behavioral: Printed Educational Handout — 12-week printed health education handout program
  Arms: Printed Health Education Materials

SUMMARY:
Sarcopenic obesity refers to a condition characterized by high body fat percentage and insufficient muscle mass, posing significant risks to physical and mental health. This issue is not limited to the elderly; it is increasingly common among younger populations as well. According to the National Nutrition and Health Survey conducted between 2017 and 2020, high rates of eating out due to study and work lifestyles in Taiwan result in limited access to nutritious food. The Ministry of Health and Welfare's statistics from 2021 show that only 33.9% of the population engages in regular exercise. Sarcopenic obesity is associated with physical activity and nutritional intake. The European Working Group on Sarcopenia in Older People has urged the public to maintain a balanced diet and establish exercise habits early to reduce the risk of sarcopenic obesity. Younger individuals are more likely to increase muscle mass with interventions in exercise and nutrition compared to older adults, making college students a key demographic for fostering healthy behaviors. Therefore, it is essential to address how to enhance their health awareness and behaviors.

Based on this, the present study aims to explore the impact of a multimedia intervention combined with a peer support model on the awareness and behaviors of college students at risk of being overweight. The research methodology involves a randomized controlled trial, participants from a medical university in central Taiwan. Body composition will be measured first, and eligible participants will be randomly assigned to either an experimental group or a control group, followed by a 12-week intervention and subsequent post-test. The study will analyze the effects of multimedia combined with peer support on the awareness and behaviors of at-risk college students, as well as assess muscle mass changes through grip strength measurements. The goal is to enhance college students' awareness of their health behaviors, improve their dietary and exercise habits, fill knowledge and application gaps, and provide an evidence-based foundation for future strategies to promote healthy behaviors among young populations.

DETAILED DESCRIPTION:
This randomized controlled trial (RCT) will recruit students from a university in central Taiwan, randomly assigning them to either an intervention or a control group.

Intervention Participants will first complete body composition assessments and questionnaires. Eligible students will be randomly assigned to the intervention or control group.

Intervention group:12-week program including weekly educational videos on exercise and nutrition.Biweekly group exercises (elastic band and aerobic).Peer support groups (5 per group) for weekly discussions and exercise tracking.

Control group:Receives weekly paper-based health education materials on exercise and diet.

Video Content Includes:

Sarcopenic Obesity Awareness: Definitions, risks, health effects, and prevention strategies.Exercise Guidance: Filmed with exercise science faculty, includes warm-up (5 min), resistance/aerobic training (20 min), and cool-down (5 min).

Nutrition Education: Based on HPA guidelines and reviewed by dietetics faculty, covering protein, vegetables, fruits, and easy dietary tips.

Data Analysis Using SPSS 25.0.Descriptive statistics and inferential analyses will be conducted.Chi-square tests (categorical data) and independent t-tests (continuous variables) will compare baseline group differences.Paired t-tests will assess within-group pre-post changes.Independent t-tests will evaluate between-group post-intervention differences.Generalized Estimating Equations (GEE) will examine time-by-group interaction effects.Statistical significance set at α < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate students in years 1 to 4 at a medical university in central Taiwan
* Body Mass Index (BMI) between 23 and 27 or body fat percentage between 25% and 35%
* Aged 18 to 25 years
* No diagnosis of any chronic disease

Exclusion Criteria:

* University students with restricted limb movement who are unable to exercise according to instructions.
* Any condition that may restrict the proper use of a dynamometer (e.g., hand pain, osteoarthritis, or rheumatoid arthritis).

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | From enrollment to the end of treatment at 12 weeks
  BMI will be calculated as weight (kg) divided by height in meters squared (m²). Measurements will be taken using the InBody 270S body composition analyzer.
  Unit of Measure: kg/m²
Body Fat Percentage Body fat mass | From enrollment to the end of treatment at 12 weeks
  Body Fat Percentage Body fat mass will be assessed using the InBody 270S. Percentage is calculated as (fat mass ÷ body weight (kg)) × 100%.
  Unit of Measure: %
Physical Activity Level (IPAQ-SF) | From enrollment to the end of treatment at 12 weeks
  Assessed using the International Physical Activity Questionnaire - Short Form (IPAQ-SF). Results expressed in MET-minutes/week. Higher scores indicate greater physical activity and better outcome.
  Unit of Measure: MET-min/week
Hand Grip Strength | From enrollment to the end of treatment at 12 weeks
  Hand grip strength measured using Jamar handheld dynamometer. Each hand is tested three times; average grip strength is recorded. Higher values indicate better strength.
  Unit of Measure: kg

CONTACTS AND LOCATIONS:
Overall Officials: Ya-Ling Tzeng, PhD, Study Director — China Medical University, Taiwan
Locations (1):
- Ya-Ling Tzeng, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No